CLINICAL TRIAL: NCT01293773
Title: Outcome of seCond Generation Drug-ELuting Stents in Patients With Diabetes Mellitus: cOmparison of Three differenT Drug Regimens
Brief Title: Outcome of Second Generation Drug-eLuting Stents in Patients With Diabetes Mellitus
Acronym: OCELOT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Policlinico Casilino ASL RMB (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Enrico Romagnoli, Policlinico Casilino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 007/CE-RMB
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Randomized controlled trial; Drug-eluting Stent; Multicenter study
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Taxus Element (Active Comparator): Patients treated with paclitaxel-eluting stent (Taxus Element, Boston Scientific, MN)
  Interventions: Device: Taxus Element stent
- Xience Prime (Active Comparator): Patients treated with Everolimus-eluting stent (Xience Prime, Abbott, IL)
  Interventions: Device: Xience Prime stent
- Integrity Resolute (Active Comparator): Patients treated with ABT 578-eluting stent (Integrity Resolute, Medtronic, MA)
  Interventions: Device: Integrity Resolute stent

INTERVENTIONS:
Device: Taxus Element stent — paclitaxel-eluting stent
  Other Names: Taxus
  Arms: Taxus Element
Device: Integrity Resolute stent — ABT 578-eluting stent
  Other Names: Resolute Integrity
  Arms: Integrity Resolute
Device: Xience Prime stent — Everolimus-eluting stent
  Other Names: Xience Prime
  Arms: Xience Prime

SUMMARY:
Design: prospective, randomized, multi-center trial comparing the safety and efficacy in the prevention of target lesion failure (TLF) of second generation paclitaxel- versus ABT578- versus Everolimus- eluting stents Study Population: all consecutive diabetic patients with de novo coronary artery lesions undergoing drug-eluting stent implantation in 2010-12.

Time Course: initial Enrollment: October 2010; end of the Enrollment: December 2012 Primary End-Point: target lesion revascularization (TLF) defined as the occurrence of cardiac death, myocardial infarction and repeated lesion revascularization within 12 months.

Secondary End-Points: 1) impact of glucose level during the first three months following the procedure (assessed by hemoglobin A1C ) on clinically-driven target lesion revascularization; 2)TLF and TLR within 12, 24 and 36 months; 3) comparison 12 months versus prolonged (> 12 months) of dual antiplatelet therapy

DETAILED DESCRIPTION:
Prospective, randomized, triple arm study. The study population will include all consecutive diabetic patients within 24 months undergoing elective second generation DES implantation for de novo coronary artery disease. In the randomization process all participating centers will be equally stratified to avoid statistical unbalance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years old
2. Presence of one or more de novo stenosis equal or greater than 70% in a native coronary artery, treated with a second generation drug-eluting stent
3. Subject and the treating physician agree that the subject will comply with all follow-up evaluations
4. Subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site

Exclusion Criteria:

1. Subject's age is < 18 years and with acute myocardial infarction in the 48 prior to the procedure
2. The patient is pregnant or breastfeeding
3. Known allergies to: aspirin, clopidogrel (Plavix) and ticlopidine (tiklid), heparin, Paclitaxel, Everolimus, ABT 578, stainless steel, or contrast agent (which cannot be adequately pre-medicated)
4. A platelet count < 75,000 cells/mm3 or > 700,000 cells/mm3 or a WBC < 3,000 cells/mm3
5. Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
6. Prior participation in this study
7. Active peptic ulcer or upper GI bleeding within the prior 3 months
8. Subject has active sepsis
9. Any lesion that is located in a saphenous vein graft
10. In the investigator's opinion, subject has a co-morbid condition(s) that could limit the life expectancy to less than one year, or limit the subject's ability to participate in the study or comply with follow-up requirements or impact the scientific integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  Target lesion failure (TLF) defined as the occurrence of cardiac death, target vessel-related myocardial infarction and repeated revascularization of the target lesion

SECONDARY OUTCOMES:
Effect of glucose levels on repeat revascularization | 1 year
  Impact of glucose level during the three months following the procedure (assessed by hemoglobin A1C ) on clinically-driven target lesion revascularization rate
Target Lesion Revascularization | 1, 2 and 3 year
  Target lesion revascularization at 12, 24 and 36 months
Effect of dual antiplatelet therapy on outcome | 3 year
  Comparison of 12-month versus prolonged (> 12-month) dual antiplatelet therapy on outcome

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Romagnoli, MD, PhD, Principal Investigator — Policlinico Casilino
Locations (2):
- Italy (2):
  - Azienda Policlinico-Universitaria di Modena, Modena, Modena
  - Policlinico Casilino, Rome, Rome